CLINICAL TRIAL: NCT00599742
Title: Comorbidity Between Balance and Childhood Anxiety: Treatment of Anxiety by Training of Balance
Brief Title: Comorbidity Between Balance and Childhood Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lev-Hasharon Mental Healtlh Center (Other Government)
Collaborators: Tel Aviv University (Other); Institute of Physical Education and Sports Sciences (Other); University of Haifa (Other)
Responsible Party: Michal Rappaport MD, Lev Hasharon Mental Health Center, Child and Adolescent Mental Health Clinic,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LH22/2007.CTIL; 920070174
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Anxiety
Keywords: Balance disorder; Vestibular disorder; Generalized anxiety disorder; Separation anxiety disorder; Children; Balance training
MeSH Terms: conditions — Anxiety Disorders; Vestibular Diseases; Generalized Anxiety Disorder; Anxiety, Separation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Balance training group
  Interventions: Behavioral: Balance training
- B (Active Comparator): Motor Training
  Interventions: Behavioral: Motor training

INTERVENTIONS:
Behavioral: Balance training — Physical exercise of balance. The training will last 7 weeks, twice per week, 1 hour per session.
  Arms: A
Behavioral: Motor training — Motor exercise of power and flexibility. The training will last 7 weeks, twice per week, 1 hour per session.
  Arms: B

SUMMARY:
Previous studies report frequent comorbidity of anxiety and sensory-motor imbalance in adults (Sklare et al., 2001). Only a few studies tested the comorbidity in children. We confirmed that: a) children with primary diagnosis of poor balance demonstrate an elevated anxiety level (Brat et al., 2006, submitted) and, b) children with primary diagnosis of generalized anxiety disorder demonstrate poor balance performance (Erez et al., 2004). These studies demonstrate the presence of balance-anxiety comorbidity in children with primary disorder of either balance or anxiety. Our theoretical reasoning formalized under the "three stage theory of learning" points to the possibility that poor balance may either predispose or cause the emergence of anxiety disorder (Erez et al., 2004). Thus, in the present study we test two predictions: (a) high prevalence of comorbidity of anxiety and balance disorders in children with a primary diagnosis of generalized or separation anxiety disorder, and, (b) intensive balance training, but not training of flexibility and power, will reduce the level of anxiety in children with primary diagnosis of anxiety.

DETAILED DESCRIPTION:
Study sample: 64 children, 8 to 14 years old, with diagnosis of generalized or separation anxiety.

Training: 32 of these children will undergo balance training and the other 32 children will undergo motor training of power and flexibility. Training will last 7 weeks, twice per week, 1 hr each session.

Tests: Balance and anxiety tests will be applied before training period, immediately after the last training session and again 2 months after the last training session.

Tests will include standard balance performance tests and questionnaires of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-14
* Boy or girl
* Generalized or separation anxiety disorder
* Agreement to participate and written informed consent

Exclusion Criteria:

* Major affective disorders
* Severe developmental disorders
* Refusal to participate

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Balance improvement and anxiety reduction | After 7 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Michal Rappaport, MD, Principal Investigator — Lev HaSharon Mental Health Center
Locations (2):
- Israel (2):
  - Child and Adolescent Mental Health Clinic, Lev Hasharon MHC, Netanya
  - Wingate Institute for Physical Education, Netanya

REFERENCES:
- [Background] Erez O, Gordon CR, Sever J, Sadeh A, Mintz M. Balance dysfunction in childhood anxiety: findings and theoretical approach. J Anxiety Disord. 2004;18(3):341-56. doi: 10.1016/S0887-6185(02)00291-8. PMID 15125981
- [Background] Sklare DA, Konrad HR, Maser JD, Jacob RG. Special issue on the interface of balance disorders and anxiety: an introduction and overview. J Anxiety Disord. 2001 Jan-Apr;15(1-2):1-7. doi: 10.1016/s0887-6185(00)00039-6. No abstract available. PMID 11388353
- See also: website of location of study — http://www.lev-hasharon.co.il